CLINICAL TRIAL: NCT02613819
Title: Focal Ablative STereotactic Radiosurgery for Cancers of the Kidney, a Phase II Clinical Trial (FASTRACK II)
Brief Title: Focal Ablative STereotactic Radiosurgery for Cancers of the Kidney
Acronym: FASTRACK II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 15.03
Record Dates: First submitted 2015-11-04; First posted 2015-11-25 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Radiotherapy;
  * Fraction schedule 1: 26Gy in 1 fraction, for tumours < 4cm in size
  * Fraction schedule 2: 42Gy in 3 fractions, for tumours > 4cm in size
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Ablative Body Radiotherapy (Experimental): Stereotactic Ablative Body Radiotherapy (SABR)
  Treatment schedule 1: 26 Gray (Gy) in 1 fraction, for tumours of less than or equal to 4cm in size.
  Treatment schedule 2: 42 Gray (Gy) in 3 fractions, for tumours of greater than 4cm in size
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — Renal cell carcinoma (RCC) is conventionally considered "radioresistant" to fully fractionated EBRT. In an effort to overcome the perceived "radioresistance" of RCC, severely hypofractionated External beam radiation therapy (EBRT) in the form of stereotactic radiotherapy will be used in the management of renal cell carcinoma with radiotherapy.
  Other Names: Stereotactic Ablative Body Radiotherapy

SUMMARY:
This study is evaluating the activity and efficacy of Stereotactic Ablative Body Radiotherapy (SABR) for the treatment of kidney cancers.

DETAILED DESCRIPTION:
Who is it for?

* Age > 18 years old
* All patients must have a biopsy confirmed diagnosis of renal cell carcinoma with a single lesion within a kidney
* ECOGperformance of 0-2 inclusive.
* Life expectancy > 9 months
* Either medically inoperable, technically high risk for surgery or decline surgery.
* Multidisciplinary decision for active treatment

Study Details:

Definitive external beam radiotherapy (EBRT) is often used to treat medically inoperable patients with cancers in many different organs, including the kidneys. However, renal cell carcinoma (RCC) is conventionally considered "radioresistant" to fully fractionated EBRT. In an effort to overcome the perceived "radioresistance" of RCC, severely hypofractionated EBRT in the form of stereotactic radiotherapy has renewed interest in the management of renal cell carcinoma with radiotherapy. This study will be evaluating the safety and effectiveness of Stereotactic Ablative Body Radiotherapy (SABR) for the treatment of cancers of the kidney.

Participants in this study will be allocated to receive either multi-fraction SABR (3 fractions over 2 weeks) or single fraction SABR (1 fraction only).

All participants will be assessed at regular intervals post treatment in order to estimate the activity and efficacy of the technique, evaluate tolerability, estimate survival, estimate distant failure rate, and renal function change after SABR.

The follow-up visits occur at 4 weeks and every 3 months in the 1st year post treatment, then every 6 months in the second year and then yearly until study closure (2 years after the last participant finishes study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* All patients must have a biopsy confirmed diagnosis of renal cell carcinoma with a single lesion within a kidney
* Eastern Cooperative Oncology Group (ECOG) performance of 0-2 inclusive.
* Life expectancy > 9 months
* Either medically inoperable, technically high risk for surgery or decline surgery.
* Multidisciplinary decision for active treatment

Exclusion Criteria:

* Pre-treatment estimated glomerular filtration rate < 30 mls/min
* Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Delivery of targeted agents (such as sunitinib) are allowable only when at least 7 days separate the delivery of the proposed agent and the delivery of the stereotactic radiotherapy.
* Previous high-dose radiotherapy to an overlapping region
* Tumours of larger than 8cm is size

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-07; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Activity and efficacy of SABR measured by Freedom from local progression assessed by RECIST Criteria | 12mths post treatment
  Responsive Evaluation Criteria in Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Tolerability of SABR Assessed as cummulative incedents of severe toxicity by CTCAE v4 | From date of treatment commencement until first documented progression or date of death from any cause, whichever came first, assessed from 4wks, 3 mths, 6 mths, 9mths, 12 mths, 18 mths, 24 mths, 33 mths, 42 mths, 51 mths, and 60 mth post treatment
  Common Terminology Criteria for Adverse Events (CTCAE)
Estimated Survival after SABR assessed by clinincal assessment | assessed up to 60 months
  Stereotactic Ablative Radiotherapy (SABR)
Estimated Distant Failure Rate after SABR assessed by CT scan and clinical assessment | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed from 6 mths, 9 mths, 12 mths, 18mths, 33 mths, 42 mths, 51 mths, and 60 mths post treatment
Renal Function Change after SABR assessed by split renal function and GFR | Baseline, 12mths post treatment, and 24 mths post treatment
  Calculated Glomular Filtration Rate (GFR)
Renal Function Change after SABR assessed by using eGFR | Baseline,3 mths, 6 mths, 9mths, 12 mths, 18 mths, 24 mths, 33 mths, 42 mths, 51 mths, and 60 mths
  Estimated Glomular Filtration Rate (eGFR)

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, A/Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Siva S, Bressel M, Sidhom M, Sridharan S, Vanneste BGL, Davey R, Montgomery R, Ruben J, Foroudi F, Higgs B, Lin C, Raman A, Hardcastle N, Hofman MS, De Abreu Lourenco R, Shaw M, Mancuso P, Moon D, Wong LM, Lawrentschuk N, Wood S, Brook NR, Kron T, Martin J, Pryor D; FASTRACK II Investigator Group. Stereotactic ablative body radiotherapy for primary kidney cancer (TROG 15.03 FASTRACK II): a non-randomised phase 2 trial. Lancet Oncol. 2024 Mar;25(3):308-316. doi: 10.1016/S1470-2045(24)00020-2. PMID 38423047
- [Derived] Siva S, Chesson B, Bressel M, Pryor D, Higgs B, Reynolds HM, Hardcastle N, Montgomery R, Vanneste B, Khoo V, Ruben J, Lau E, Hofman MS, De Abreu Lourenco R, Sridharan S, Brook NR, Martin J, Lawrentschuk N, Kron T, Foroudi F. TROG 15.03 phase II clinical trial of Focal Ablative STereotactic Radiosurgery for Cancers of the Kidney - FASTRACK II. BMC Cancer. 2018 Oct 23;18(1):1030. doi: 10.1186/s12885-018-4916-2. PMID 30352550